CLINICAL TRIAL: NCT06876116
Title: Comparison of Therapeutic Effects of Once-daily Fluorometholone 0.1% Versus Twice-daily Cyclosporine 0.05% in Patients With Dry Eye Disease: A Randomized, Assessor-blinded Clinical Trial
Brief Title: Once-daily Fluorometholone vs Twice-daily Cyclosporine in Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dong Hyun Kim, Principal Investigator, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022AN0569
Record Dates: First submitted 2025-02-25; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Fluorometholone; Ophthalmic Solutions; Cyclosporine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- once-daily fluorometholone 0.1% group (Active Comparator): After induction therapy with fluorometholone 0.1% four times a day for 4 weeks, patients continued with fluorometholone 0.1% once a day for 8 weeks.
  Interventions: Drug: Fluorometholone 0.1% ophthalmic solution
- twice-daily cyclosporine 0.05% group (Active Comparator): After induction therapy with fluorometholone 0.1% four times a day for 4 weeks, patients continued with cyclosporine 0.05% twice a day for 8 weeks.
  Interventions: Drug: Cyclosporine 0.05% eye drops

INTERVENTIONS:
Drug: Fluorometholone 0.1% ophthalmic solution — After induction therapy with fluorometholone 0.1% four times a day for 4 weeks, patients continued with fluorometholone 0.1% once a day for 8 weeks.
  Arms: once-daily fluorometholone 0.1% group
Drug: Cyclosporine 0.05% eye drops — After induction therapy with fluorometholone 0.1% four times a day for 4 weeks, patients continued with cyclosporine 0.05% twice a day for 8 weeks.
  Other Names: fluorometholone 0.1%
  Arms: twice-daily cyclosporine 0.05% group

SUMMARY:
This study compares the therapeutic effects of once-daily fluorometholone 0.1% versus twice-daily cyclosporine 0.05% after short-term fluorometholone induction treatment in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. participants aged 18 years or older
2. complaint of dry eye symptoms for 6 months or longer at screening
3. ocular surface disease index (OSDI) score of 33 or higher
4. tear film breakup time of 7 seconds or less

Exclusion Criteria:

1. abnormal lid anatomy or active blepharitis
2. severe systemic autoimmune diseases
3. received permanent lacrimal plug within 3 months
4. DED secondary to alkali burns, cicatricial pemphigoid, or Stevens-Johnson syndrome
5. ocular/periocular malignancy
6. active ocular allergies or allergy to the study drug or its components
7. active infection
8. intraocular surgery or ocular laser surgery within 6 months
9. uncontrolled systemic disease or history of herpetic keratitis
10. contact lens user
11. intraocular pressure >25mmHg
12. pregnancy or current breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) score | From enrollment to the end of treatment at 12 weeks
  Score 0-100
tear breakup time (TBUT) | From enrollment to the end of treatment at 12 weeks
  Unit: Seconds
corneal staining score (CSS) | From enrollment to the end of treatment at 12 weeks
  National Eye Institute Scale, 0-15
Schirmer's test | From enrollment to the end of treatment at 12 weeks
  Unit: mm/5 min
Meibomian gland dysfunction grade (0-4) | From enrollment to the end of treatment at 12 weeks
  Scale 0-4
tear matrix metalloproteinase-9 (MMP-9) grade | From enrollment to the end of treatment at 12 weeks
  Grade 0-4
tear osmolarity | From enrollment to the end of treatment at 12 weeks
  Unit: mOsm/L

SECONDARY OUTCOMES:
Tear IL-6 levels | From enrollment to the end of treatment at 12 weeks
  Unit: pg/mL
tear 8-oxo-dG levels | From enrollment to the end of treatment at 12 weeks
  Unit: pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not openly available due to reasons of sensitivity and may available from the corresponding author upon reasonable request.